CLINICAL TRIAL: NCT06089538
Title: Electrophysiological Signatures of Cognitive Disorders Related to ICU Delirium : a Pilot Study
Brief Title: Electrophysiological Signatures of Cognitive Disorders Related to Intensive Care Unit (ICU) delirium_ BRAINSTORM-EEG
Acronym: B-EEG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC31/22/0526; 2023-A00935-40 (Other: ID-RCB)
Record Dates: First submitted 2023-09-13; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Cognitive Dysfunction
Keywords: delirium; acute respiratory distress syndrome (ARDS); P300; N400; self-processing; semantic priming; functional connectivity
MeSH Terms: conditions — Cognitive Dysfunction; Delirium; Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Delirium patients group (Experimental): Patients admitted for acute respiratory distress syndrome (ARDS) who developed delirium
  Interventions: Diagnostic Test: mEEG battery
- Patients without delirium (Active Comparator): Patients admitted for acute respiratory distress syndrome (ARDS) who did not developed delirium
  Interventions: Diagnostic Test: mEEG battery

INTERVENTIONS:
Diagnostic Test: mEEG battery — The 2 groups will be assessed twice : in the acute phase of acute respiratory distress syndrome (ARDS) at patient's bedside in the intensive care unit (ICU) using an mEEG battery (electrophysiological acquisition at rest and during complex cognitive stimulation), and a simple clinical neuropsychological assessment ; 6 months ± 2 weeks later using the same mEEG battery and a multi-domain clinical neurocognitive and psychological assessment battery

SUMMARY:
Early cognitive assessment of critically-ill acute respiratory distress syndrome (ARDS) patients with delirium using a multidimensional electrophysiological evaluation battery (mEEG) to identify and characterize the neural correlates of cognitive dysfunctions associated with delirium (vigilance, attention, semantic and lexical processing, self-processing), and to develop a prognostic evaluation of neurocognitive and psychological disorders using an innovative non-behavioral approach.

DETAILED DESCRIPTION:
Delirium is an altered mental status associated with specific manifestations such as reduced ability to direct, focus, maintain and shift attention Diagnostic Medical Systems V criteria (DSM). The vulnerability of critically-ill acute respiratory distress syndrome (ARDS) patients explains the high incidence of delirium (up to 80%) in this setting. Delirium is an independent predictor of post-traumatic stress disorder, long term cognitive decline and mortality. To reduce this medical and social burden, a more complete description of delirium is needed both in terms of cognitive impairments and long term neurological and neuropsychological impact. Actually, it could be argued that the current exclusive behavioral assessment of these patients is insufficient in terms of diagnosis and prognostic assessment. In recent years, the study of consciousness has made major progress thanks to the use of innovative electrophysiological exploration methods. This work has notably allowed the development of new non-behavioral tools for the exploration of brain function in brain damaged patients in response to complex auditory stimulations (multidimensional electrophysiological battery, mEEG). In this context, the investigators have recently demonstrated alterations in cognitive functions related to language- and self-processing in acute respiratory distress syndrome (ARDS) patients with severe acute respiratory syndrome (SARS) - COVID-19 infection. These electrophysiological cognitive alterations were particularly marked in COVID-19 patients with delirium. Further studies are needed to disentangle the cognitive impact specifically related to delirium from that related to a severe form of COVID-19. The primary objective of this study is to identify diagnostic electrophysiological signatures of cognitive dysfunctions associated with the acute phase of delirium in critically-ill acute respiratory distress syndrome (ARDS) patients using a multidimensional electrophysiological assessment (mEEG) recording at rest and during auditory stimulation (first visit). Secondary objectives are to characterize the impact of intensive care unit (ICU)-related delirium on neurocognitive and psychological dysfunctions observed at 6 months (second visit), in order to explore the prognostic predictive value of electrophysiological data acquired during the acute phase of delirium.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the intensive care unit with ARDS (according to Berlin criteria)
* Membership of a social security scheme
* Signed consent of the patient (group without delirium) or referring person (group with delirium)
* Discontinuation of any sedative agent for ≥ 72 hours

Exclusion Criteria:

* Pre-existing psychotic disorders
* Pre-existing cognitive deficits
* Patients with chronic ethylism
* Previous neurological history
* Recent ICU admission (> 5 days of ICU hospitalization within 6 months prior to current ICU admission)
* Patients whose delirium cannot be reliably assessed due to blindness, deafness or inability to speak French
* Patients whose life expectancy is unlikely to exceed 24 hours
* Pregnant women
* Patients under court protection
* Patients who have already participated in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-30 (Estimated); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-06-20 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of the signal of weighted Symbolic Mutual Information (wSMI) measured by multidimensional ElectroEncephaloGram (mEEG) at the acute phase of delirium | Baseline
  Analysis of data from the multidimensional electrophysiological battery (mEEG) at the acute phase of delirium: weighted Symbolic Mutual Information (wSMI) measured by presence or absence of the signal
Amplitude of the signal of weighted Symbolic Mutual Information (wSMI) measured by multidimensional ElectroEncephaloGram (mEEG) at the acute phase of delirium | Baseline
  Analysis of data from the multidimensional electrophysiological battery (mEEG) at the acute phase of delirium: weighted Symbolic Mutual Information (wSMI) measured by amplitude (microvolts)
Latency of the signal of weighted Symbolic Mutual Information (wSMI) measured by multidimensional ElectroEncephaloGram (mEEG) at the acute phase of delirium | Baseline
  Analysis of data from the multidimensional electrophysiological battery (mEEG) at the acute phase of delirium: weighted Symbolic Mutual Information (wSMI) measured by latency (milliseconds)
Presence or absence of the signal of weighted Symbolic Mutual Information (wSMI) measured by multidimensional ElectroEncephaloGram (mEEG) six months after phase of delirium | 6 months
  Analysis of data from the multidimensional electrophysiological battery (mEEG) six months after phase of delirium: weighted Symbolic Mutual Information (wSMI) measured by presence or absence of the signal
Amplitude of the signal of weighted Symbolic Mutual Information (wSMI) measured by multidimensional ElectroEncephaloGram (mEEG) at the acute phase of delirium | 6 months
  Analysis of data from the multidimensional electrophysiological battery (mEEG) six months after phase of delirium: weighted Symbolic Mutual Information (wSMI) measured by amplitude (microvolts)
Latency of the signal of weighted Symbolic Mutual Information (wSMI) measured by multidimensional ElectroEncephaloGram (mEEG) at the acute phase of delirium | 6 months
  Analysis of data from the multidimensional electrophysiological battery (mEEG) six months after phase of delirium: weighted Symbolic Mutual Information (wSMI) measured by latency (milliseconds)

CONTACTS AND LOCATIONS:
Overall Officials: William BUFFIERES, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital of Toulouse, Toulouse, France